CLINICAL TRIAL: NCT07301957
Title: Impact of Early Rupture of the Residual Membrane on Latency Before Labour Begins
Acronym: RESIRUPT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHM-2023/S30/07
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Prelabor Rupture of Membranes
Keywords: prelabor rupture of membranes
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional rupture of the residual membrane (Experimental): Rupture of the residual membrane
  Interventions: Other: Additional rupture of the residual membrane
- Standard of care (No Intervention): unbroken residual membrane

INTERVENTIONS:
Other: Additional rupture of the residual membrane — Additional rupture of the residual membrane using a sterile, single-use amniotic membrane piercer such as the Robé device
  Arms: Additional rupture of the residual membrane

SUMMARY:
Approximately 25% of patients experience premature rupture of membranes before labour. Of these patients, 82% will give birth within 24 hours and 97% within 48 hours.

Patients who do not go into labour spontaneously will be induced 24 or 48 hours after their membranes rupture, depending on the centre.

During this period, they are hospitalised in the obstetrics department. The presence of a residual membrane appears to prolong the latency period before labour begins and the rate of induction, according to a pilot study conducted by investigator.

No study specifically addresses this topic. The various studies on "Rupture of Membranes Before Labour" assess its frequency of occurrence or the time before considering induction. They also assess the occurrence of maternal-foetal infection. This is no longer of interest today, as antibiotic prophylaxis has significantly reduced maternal-foetal infections.

Investigator would therefore like to assess the impact of additional rupture of the residual membrane upon the patient's admission on the latency before labour and the induction rate (for membrane rupture exceeding 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Single foetal pregnancy, cephalic presentation
* diagnosis of membrane rupture with persistence of one membrane and absence of immediate spontaneous labour.
* Person affiliated with or beneficiary of a social security scheme
* Free, informed and written consent signed by the participant and the investigator (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Minor patient
* patient under guardianship/curatorship,
* multiple pregnancy, pregnancy with foetal death
* non-cephalic presentation
* gestational age less than 37 weeks,
* rupture of membranes more than 12 hours ago
* contraindication to vaginal deliver
* meconium-stained amniotic fluid,
* clinical signs suggestive of intrauterine infection (maternal hyperthermia >38°C, maternal and/or foetal tachycardia, purulent amniotic fluid),
* cervix not accessible for artificial rupture
* vaginismus
* contraindication to a potential expectant management
* indication for induction for another reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Latency between the rupture of membranes and the onset of labour | At labour onset (up to 6 days)
  Latency is evaluated by the time in minutes between the rupture of membranes and the onset of labour. The diagnosis of rupture is the spontaneous loss of fluid through the vagina. The diagnosis of labour is defined by the onset of painful uterine contractions and cervical changes. The time recorded will be when the patient's cervix is 3 cm dilated.

SECONDARY OUTCOMES:
Trigger rate for prolonged rupture of membranes | 48 hours after rupture of membranes
  Trigger rate for prolonged rupture of membranes was evaluated by absence of spontaneous labour 48 hours after the time H0 defined during the initial consultation (rupture of membrane's diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Charlotte FAURANT, MD, Principal Investigator — Centre Hospitalier le Mans
Locations (2):
- France (2):
  - CHU Angers, Angers
  - Centre Hospitalier Le Mans, Le Mans